CLINICAL TRIAL: NCT05205473
Title: Sciatic Nerve Blockade by Subgluteal Access 12.5 ml of 1% Lidocaine: US Guidance Versus US Guidance With Electrical Stimulation of Peripheral Nerves (Influence of the Sciatic Nerve Blockade on the Effectiveness of Small Doses of Local Anesthetic.).
Acronym: EPBwEPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mogilev Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Valery Piacherski, Ph.D., Chief of the Department of Anesthesiology and Intensive Care, Mogilev Regional Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12.5ml sciatic nerve
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Nerve Block; Efficiency; Sciatic Nerve; Ultrasonography; Minimum Effective Dose
Keywords: sciatic nerve block; ultrasound guidance; electrical stimulation of peripheral nerves; lidocaine; Аnesthetics Local; Minimum Effective Dose
MeSH Terms: interventions — Lidocaine; Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SN blockade under ultrasound control with a peripheral nerve stimulator 12.5 ml 1% lidocaine (Active Comparator): Patients undergoing surgery on the knee, shin, ankle or foot
  Interventions: Procedure: Sciatic nerve block under ultrasound control with a electrostimulator peripheral nerves 12.5 ml 1% lidocaine
- SN blockade under ultrasound control without a peripheral nerve stimulator (Experimental): Patients undergoing surgery on the knee, shin, ankle or foot
  Interventions: Procedure: sciatic nerve blockade under ultrasound control without a peripheral nerve stimulator 12.5 ml 1% lidocaine

INTERVENTIONS:
Procedure: Sciatic nerve block under ultrasound control with a electrostimulator peripheral nerves 12.5 ml 1% lidocaine — Following the ultrasound visualization of the femoral nerve, a insulated injection needle was connected to the nerve stimulator . Under ultrasound visualization guidance, the needle of the electronic nerve stimulator was positioned at the sciatic nerve (in plane) from its lateral side at a slightly superior position . A marker for LA introduction was the visualization of the needle end near the nerve, and a positive muscular response . Subsequently, the introduction of LA solution was initiated (12.5 ml 1% lidocaine).If LA was spreading from the lateral side down to the nerve, then the needle was replaced to the upper point of the nerve and the rest of LA was introduced, and vice versa . The presence of a complete and incomplete spread of LA along the entire circumference of the nerve was assessed. Correspondingly, if the anesthetic was spreading upwardly, the needle would be downwardly replaced.
  In addition, a femoral nerve block is performed.
  Other Names: Anesthesia for lower limb surgery
  Arms: SN blockade under ultrasound control with a peripheral nerve stimulator 12.5 ml 1% lidocaine
Procedure: sciatic nerve blockade under ultrasound control without a peripheral nerve stimulator 12.5 ml 1% lidocaine — Under ultrasound visualization guidance, the needle owas positioned at the sciatic nerve (in plane) from its lateral side at a slightly superior position . A marker for LA introduction was the visualization of the needle end near the nerve. Subsequently, the introduction of LA solution was initiated. The position of the needle was corrected 1-2 times according to the type of anesthetic spread. If LA was spreading from the lateral side down to the nerve, then the needle was replaced to the upper point of the nerve and the rest of LA was introduced, and vice versa . The presence of a complete and incomplete spread of LA (12.5 ml 1% lidocaine) along the entire circumference of the nerve was assessed. Correspondingly, if the anesthetic was spreading upwardly, the needle would be downwardly replaced.
  In addition, a femoral nerve block is performed.
  Other Names: Anesthesia for lower limb surgery
  Arms: SN blockade under ultrasound control without a peripheral nerve stimulator

SUMMARY:
In modern anesthesiology, peripheral nerve blocks are performed using ultrasound control and electrical stimulation of peripheral nerves (PEN), or only ultrasound control or only EPN. The most effective methods are with the use of ultrasound control. Until now, the effectiveness of the sciatic nerve blockade by the subgluteal approach, performed only under ultrasound control without EPN, in comparison with the blockade of the sciatic nerve performed under ultrasound control with EPN, has not been established.

There is no data on how the effectiveness of the blockade of the sciatic nerve with small doses of lidocaine is influenced by the method of performing the blockade: under ultrasound control versus ultrasound control with electrostimulation of the nerve.

Research hypothesis: the blockade of the sciatic nerve by the subgluteal approach (12.5 ml 1%lidocaine -Minimum Effective Dose - previously established ) performed only under ultrasound control has the same effectiveness as the blockade performed under the ultrasound control with EPN.

ELIGIBILITY:
Inclusion Criteria:

* indication requiring anesthesia maintenance;
* patient's written consent about the type of anesthesia and possible complications of regional anesthesia

Exclusion Criteria:

* patient's refusal of application for the proposed form of anesthesia;
* patients younger than 18 years;
* patients weighing less than 50 kg;
* a physical status score of more than 3 determined by the American Society of Anesthesiologists (ASA);
* a history of allergic reactions to the drugs used;
* coagulopathies;
* infections of the skin at the injection site;
* neurological or neuromuscular diseases;
* severe liver diseases or kidney failures;
* an inability to cooperate with the patient.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Сomplete sensory sciatic nerve block | The quality of sensory blocks was assessed after 45 min of administration of the sciatic nerve block. The evaluation of the block was carried out by an anesthesiologist who was not involved in the study, and was blinded to solution that had been
  The stimulus of the needle prick was applied to check the sensory block of the sciatic nerve. Stimulation with a needle is carried out in the area of innervation of the sciatic nerve below the knee The assessment of skin sensitivity was carried out with the help of a similar scale: + +\ indicating a complete sensory block; +\ indicating a partial sensory block, a patient was unable to differentiate between the type of stimuli ; and -\ indicating that the skin sensitivity was fully preserved.
Сomplete motor sciatic nerve block | The quality of motor blocks was assessed after 45 min of administration of the sciatic nerve block. The evaluation of the block was carried out by an anesthesiologist who was not involved in the study, and was blinded to solution that had been
  The assessment of the motor block was carried out with the help of the following scale: + +\ which indicated that movements were completely absent; +\ which indicated that movements were partially preserved or were uncoordinated; and -\ which indicated that movements were fully preserved.Flexion-extension of the foot and toes is assessed
The need for additional pain relief during surgery | During the operation (start of operation - end of operation)
  The need for additional use of narcotic analgesics or local anesthesia during surgery (criterion-reporting of painful feelings during the operation). Based on the patient's complaint about pain of any intensity during the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Valery Piacherski, Principal Investigator — Mogilev Regional Clinical Hospital; Lidziya Muzyka, Principal Investigator — Mogilev Regional Clinical Hospital
Locations (1):
- Mogilev Regional Clinical Hospital, Mogilev, Belarus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publishing the data
Access Criteria: Contact us: Valery Piacherski, Ph.D.; pechersky.v@yandex.ru